CLINICAL TRIAL: NCT05805345
Title: Clinical Comparison of Toric Contact Lenses Fit Characteristics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLF993-P001
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Astigmatism; Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Astigmatism; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- DT1fA/T30fA/AOHGfA/P1fA (Other): DT1fA worn first, followed by T30fA, as randomized, during the first wear period, with AOHGfA worn first, followed by P1fA during the second wear period. Each lens type will be worn in both eyes for approximately 30 minutes. The wear periods will be separated by 1 to 9 days.
  Interventions: Device: Delefilcon A toric soft contact lens; Device: Lehfilcon A toric soft contact lens; Device: Lotrafilcon B toric soft contact lens; Device: Verofilcon A toric soft contact lens
- T30fA/AOHGfA/P1fA/DT1fA (Other): T30fA worn first, followed by AOHGfA, as randomized, during the first wear period, with P1fA worn first, followed by DT1fA during the second wear period. Each lens type will be worn in both eyes for approximately 30 minutes. The wear periods will be separated by 1 to 9 days.
  Interventions: Device: Delefilcon A toric soft contact lens; Device: Lehfilcon A toric soft contact lens; Device: Lotrafilcon B toric soft contact lens; Device: Verofilcon A toric soft contact lens
- AOHGfA/P1fA/DT1fA/T30fA (Other): AOHGfA worn first, followed by P1fA, as randomized, during the first wear period, with DT1fA worn first, followed by T30fA during the second wear period. Each lens type will be worn in both eyes for approximately 30 minutes. The wear periods will be separated by 1 to 9 days.
  Interventions: Device: Delefilcon A toric soft contact lens; Device: Lehfilcon A toric soft contact lens; Device: Lotrafilcon B toric soft contact lens; Device: Verofilcon A toric soft contact lens
- P1fA/DT1fA/T30fA/AOHGfA (Other): P1fA worn first, followed by DT1fA, as randomized, during the first wear period, with T30fA worn first, followed by AOHGfA during the second wear period. Each lens type will be worn in both eyes for approximately 30 minutes. The wear periods will be separated by 1 to 9 days.
  Interventions: Device: Delefilcon A toric soft contact lens; Device: Lehfilcon A toric soft contact lens; Device: Lotrafilcon B toric soft contact lens; Device: Verofilcon A toric soft contact lens

INTERVENTIONS:
Device: Delefilcon A toric soft contact lens — Commercially available silicone hydrogel contact lens
  Other Names: DT1fA; DAILIES TOTAL1® for Astigmatism
Device: Lehfilcon A toric soft contact lens — Commercially available silicone hydrogel contact lens
  Other Names: T30fA; TOTAL30™ for Astigmatism
Device: Lotrafilcon B toric soft contact lens — Commercially available silicone hydrogel contact lens
  Other Names: AOHGfA; AIR OPTIX® plus HydraGlyde® for Astigmatism
Device: Verofilcon A toric soft contact lens — Commercially available silicone hydrogel contact lens
  Other Names: P1fA; PRECISION1® for Astigmatism

SUMMARY:
The purpose of this study is to compare the fit characteristics between four Alcon commercially available toric contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 visits including the screening visit. The total duration of a subject's participation in the study will be approximately 19 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of toric soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Able to be fit with contact lenses within the available range of sphere, cylinder power, and axes (based on lens availability).
* Best Corrected Visual Acuity (BCVA) better than or equal to 0.10 (logMAR) in each eye.
* Willing to stop wearing habitual contact lenses during in-office visits.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current spherical, monovision or multifocal lens wearer.
* Protocol-specified biomicroscopy findings at screening.
* Current or history of herpetic keratitis in either eye.
* Participation in a clinical trial within the previous 30 days or currently enrolled in any clinical trial.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Distance VA with study lenses | 30 mins (± 15 mins), each product
  Visual Acuity (VA) will be assessed using letter charts with study lenses in place and reported in logarithm minimum angle of resolution (logMAR). A logMAR value of 0.0 equates to 20/20 Snellen, which is considered normal distance eyesight. Eyes will be assessed individually.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Chair — Alcon Research, LLC
Locations (7):
- United States (7):
  - Kurata Eyecare Center, Los Angeles, California
  - Omega Vision Center P.A., Longwood, Florida
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Kannarr Eye Care LLC, Pittsburg, Kansas
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee
  - Clarke EyeCare Center, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No